CLINICAL TRIAL: NCT01858870
Title: Observational Retrospective Study of Effectivity and Tolerability in Patients With Lacosamide Medication
Status: Completed | Type: Observational
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Other Study IDs: LACO-EXP
Record Dates: First submitted 2013-05-13; First posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2012-12

CONDITIONS: Epilepsy
Keywords: Lacosamide; Partial Crisis
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Lacosamide: patients with Partial Crisis of epilepsy treated with Lacosamide for at least 12 months
  Interventions: Drug: lacosamide

INTERVENTIONS:
Drug: lacosamide — routine clinical practice
  Other Names: Vimpat 50mg; 100mg; 150mg; 200mg

SUMMARY:
Lacosamide is an antiepileptic drug approved for using like adjuvant treatment in adults epileptic crisis.

Previous studies has granted to the adjuvant therapy a significant efficacy. This is an observational study, multicenter and retrospective, in patients with epilepsy. The aim of study is the evaluation of the adjuvant treatment with Lacosamide administered over 12 months.

The investigators will collect information from 860 patients in 13 spanish centers.

The secondary aim is assess the tolerability of treatment during 3,6 and 12 month.

DETAILED DESCRIPTION:
During the treatment we will performed a analysis in three different times (3, 6 and 12 month)for obtain a vision of tolerability and efficacy for Lacosamide in usual clinical practice. We intended describe the differences when we add Lacosamide to an antiepileptic drug, sodium channel blocker or no-sodium channel blocker in usual clinical practice.

Clinical data obtained through post-hoc analysis for registered pivotal studies made in highly refractory epileptic patients show that adjuvant treatment with Lacosamide has an extra efficacy compared with placebo. It is self-depended to the treatment with or without sodium channel blockers.

This study will allow us to obtain information about real existing most population where do not exist as high refractoriness as the pivotal studies.

The population of study is:

Patients with epilepsy, with plus that 18 years old patients, with initial partial crisis treated with Lacosamide according to usual clinical practice in Spain.

Lacosamide must has been used for epilepsy treatment at least during 12 month.

The data record is collection in 5 months.

Inclusion criteria:

1. Adults (+18).
2. Patients with epilepsy partial crisis diagnostic that had been treated with Lacosamide according to usual clinical practice.
3. The patient had at least one partial crisis during the year before to the initiation of treatment with Lacosamide.
4. The patient or their legal agent is reliable and is be able to adhere to the protocol according to the investigation criteria.

Exclusion criteria:

1. Patient is in an other study of medical protocol or medical implant.
2. Patients with other kind of epilepsy.
3. patients with chronic alcoholism or abuse drug recording in the last year.
4. patients who don't be in possession of their faculties in the moment to sign Informed Consent.

ELIGIBILITY:
Inclusion Criteria:

1. The patient, male or female, over 18 years.
2. The patient has a diagnosis of prostate cancer of any kind, and has been treated with Lacosamide according to routine clinical practice.
3. The patient had at least one Partial Crisis during the year prior to initiation of treatment with Lacosamide.
4. The patient or their legal representative is reliable and able to adhere to the protocol (ie, is able to understand and complete the interview at the study visit), at the discretion of the investigator.

Exclusion Criteria:

1. Patient is participating in another study of a medicinal product research (PMI) or a medical implant.
2. Patients with other types of epilepsy.
3. Patients with a history of chronic alcoholism or drug abuse in the last year.
4. Patients who are not in possession of his faculties at the time of obtaining the Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is designed to collect data from patients with epilepsy, aged 18 years with partial onset seizures (Partial Crisis) treated with Lacosamide as routine clinical practice in Spain. Lacosamide must have been used for the treatment of Partial Crisis for at least 12 months. We intend to collect data from approximately 860 patients in 13 Spanish centers.
Sampling Method: Probability Sample
Enrollment: 860 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The percentage of responders (patients with a crisis reduction of> 50%) at 12 months of treatment. | twelve months
  The primary objective of the study is to assess the efficacy of through in patients with Partial Crisis, with a minimum duration of 12 months.

SECONDARY OUTCOMES:
Percentage of patients reporting Adverse Events spontaneously potentially caused by the drug. | twelve months
  The secondary objective is to assess the tolerability of treatment with through in patients with Partial Crisis at 3, 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Vicente V Villanueva, doctor, Principal Investigator — Iis la Fe
Locations (1):
- Iis la Fe, Valencia, Valencia, Spain